CLINICAL TRIAL: NCT04313153
Title: Phase 3b, Randomized, Open-label, Active-controlled Trial Evaluating the Efficacy and Safety of Oral Vadadustat Once Daily (QD) and Three Times Weekly (TIW) for the Maintenance Treatment of Anemia in Hemodialysis Subjects Converting From Erythropoiesis-Stimulating Agents (ESAs)
Brief Title: Trial Evaluating the Efficacy and Safety of Oral Vadadustat Once Daily (QD) and Three Times Weekly (TIW) for the Maintenance Treatment of Anemia in Hemodialysis Subjects Converting From Erythropoiesis-Stimulating Agents (ESAs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 404-201-00012; AKB-6548-CI-0036 (Other: Akebia Protocol Number); 2019-004851-36 (EudraCT Number)
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Anemia
Keywords: vadadustat; hemodialysis; erythropoiesis-stimulating agents; darbepoetin alfa; CKD; Anemia
MeSH Terms: conditions — Anemia | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Masking Description: This is an open-label, Sponsor-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vadadustat once daily (QD) (Experimental)
  Interventions: Drug: Vadadustat
- Vadadustat three times weekly (TIW) (Experimental)
  Interventions: Drug: Vadadustat
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Vadadustat — oral tablets
  Arms: Vadadustat once daily (QD); Vadadustat three times weekly (TIW)
Drug: Darbepoetin alfa — intravenous or subcutaneous solution
  Arms: Darbepoetin alfa

SUMMARY:
This trial will be conducted to demonstrate the efficacy and safety of vadadustat compared to darbepoetin alfa for the maintenance treatment of anemia in hemodialysis participants after conversion from current erythropoiesis-stimulating agent (ESA) therapy.

DETAILED DESCRIPTION:
This study consists of three periods:

1. Screening Period
2. Conversion and Maintenance Treatment Period
3. Safety Follow-up Period

Individual participants will participate in total trial duration of approximately 64 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chronic, outpatient three times weekly (TIW) in-center hemodialysis for end-stage renal disease for at least 12 weeks prior to Screening
* Hemodialysis adequacy as indicated by single-pool Kt/Vurea ≥ 1.2 using the most recent historical measurement within 8 weeks prior to or during Screening
* Use of any approved erythropoiesis-stimulating agents (ESAs) for at least the 8 weeks prior to Screening Visit 2
* Two hemoglobin (Hb) values, at least 4 days apart, measured by the central laboratory during Screening within the following prespecified ranges:

  1. Hb values between 8.0 and 11.0 grams per deciliter (g/dL) (inclusive) in the United States;
  2. Hb values between 9.0 and 12.0 g/dL (inclusive) in Europe
* Serum ferritin ≥ 100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥ 20% during Screening
* Folate and vitamin B12 measurements ≥ lower limit of normal during Screening

Exclusion Criteria:

* Anemia due to a cause other than chronic kidney disease (e.g., sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia)
* Participants meeting cut-off of the following equivalent mean weekly doses calculated over 8 weeks prior to Screening Visit 2

  1. Methoxy polyethylene glycol-epoetin beta > 50 micrograms (µg)/week;
  2. Darbepoetin alfa > 100 µg/week;
  3. Epoetin analogues > 23000 International Units (IU)/week
* Active bleeding or recent blood loss within 8 weeks prior to randomization
* Red blood cell transfusion within 8 weeks prior to randomization
* Current uncontrolled hypertension.
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure (HF) or New York Heart Association Class IV HF, or stroke within 12 weeks prior to or during Screening.
* Known hypersensitivity to vadadustat, darbepoetin alfa, or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (54):
- United States (34):
  - Research Site, Chula Vista, California
  - Research Site, Granada Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Northridge, California
  - Research Site, San Dimas, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, Middlebury, Connecticut
  - Research Site, Coral Gables, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Pontiac, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Brookhaven, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Durham, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Hampton, Virginia
- Czechia (6):
  - Research Site, Mariánské Lázně
  - Research Site, Nový Jičín
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Slaný
- Hungary (5):
  - Research Site, Baja
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Pécs
- Italy (2):
  - Research Site, Pavia
  - Research Site, Vicenza
- Poland (5):
  - Research Site, Biała Podlaska
  - Research Site, Brodnica
  - Research Site, Lodz
  - Research Site, Pszczyna
  - Research Site, Sochaczew
- Spain (2):
  - Research Site #2, Barcelona
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kooienga L, Burke S, Kathresal A, Luo W, Yang Z, Zhang Z, Zwiech R, Hernandez GT. Safety and Efficacy of Vadadustat Once Daily and Three Times Weekly in Patients With Dialysis-Dependent CKD With Anemia. Kidney360. 2024 Nov 1;5(11):1652-1661. doi: 10.34067/KID.0000000567. Epub 2024 Sep 4. PMID 39231617
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open-label, active-controlled study of vadadustat versus darbepoetin alfa for the maintenance treatment of anemia in hemodialysis participants, after conversion from erythropoiesis-stimulating agent (ESA therapy).
Pre-assignment Details: A total of 319 participants were enrolled in the study. Data was collected by the arm to which participants were randomized and not by dose received in vadadustat QD or vadadustat TIW arms.
Groups:
- Vadadustat QD: Participants were randomized to receive vadadustat QD orally. Vadadustat starting daily dose was determined by pre-Baseline mean weekly darbepoetin alfa dose (or ESA equivalent). In the low darbepoetin alfa dose group (less than or equal to [<=] 0.45 micrograms per kilograms per week [mcg/kg/week]), participants received an initial vadadustat daily dose of 300 milligrams (mg) daily. In the high darbepoetin alfa dose group (> 0.45 and <= 1.5 mcg/kg/week), participants received an initial vadadustat daily dose of 450 mg daily. Vadadustat was titrated to achieve and maintain target hemoglobin (Hb) levels. The dose range for titration was 150 to 900 mg vadadustat QD.
- Vadadustat TIW: Participants were randomized to receive vadadustat TIW orally. Vadadustat starting daily dose was determined by pre-Baseline mean weekly darbepoetin alfa dose (or ESA equivalent). In the low darbepoetin alfa dose group (<= 0.45 mcg/kg/week), participants received an initial vadadustat dose of 600 mg TIW. In the high darbepoetin alfa dose group (> 0.45 and <= 1.5 mcg/kg/week), participants received an initial vadadustat dose of 750 mg TIW. Vadadustat was titrated to achieve and maintain target Hb levels. The dose range for titration was 150 to 1200 mg vadadustat TIW.
- Darbepoetin Alfa: Participants were randomized to receive darbepoetin alfa as a solution in single-dose prefilled syringes via intravenous (IV) injection through dialysis vascular access. For participants who had received darbepoetin alfa during screening, the initial dosing regimen was approximately the same weekly dose that they were receiving prior to randomization. For participants who had received darbepoetin alfa for the first time, the initial dosing regimen was determined by the United States Package Insert (USPI) or European Union Summary of product characteristics (EU SmPC), per the medical judgment of the investigator.
Period: Overall Study
Arm/Group | Vadadustat QD | Vadadustat TIW | Darbepoetin Alfa
Started (Randomized Population is defined as all participants who were randomized in the study have been presented in Participant Flow) | 105 | 106 | 108
Completed | 54 | 50 | 67
Not Completed | 51 | 56 | 41
Not completed — Adverse Event (includes Death) | 14 | 19 | 10
Not completed — Physician Decision | 4 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 2
Not completed — Lack of Efficacy | 3 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Receipt of a Solid Organ, Hematopoietic Stem Cell, or Bone Marrow Transplantation | 0 | 2 | 3
Not completed — Meeting Criteria for Trial Medication Stopping Rules | 16 | 20 | 19
Not completed — Change in Dialysis Modality | 0 | 1 | 2
Not completed — Permanent Change in Frequency of In-center Hemodialysis from TIW | 1 | 0 | 0
Not completed — Other | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Population is defined as all participants randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat QD | Vadadustat TIW | Darbepoetin Alfa | Total
Number analyzed (Participants) | 105 | 106 | 108 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.4) | 61.2 (12.5) | 60.8 (12.8) | 61.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 43 | 136
  Male | 58 | 60 | 65 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 36 | 26 | 85
  Not Hispanic or Latino | 82 | 70 | 82 | 234
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 4 | 1 | 3 | 8
  Black Or African American | 31 | 30 | 33 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 1 | 3
  White | 68 | 67 | 71 | 206
  Not Reported | 1 | 3 | 0 | 4
  Reported as Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hb to the Average Over the Primary Evaluation Period (PEP) (Weeks 20 to 26)
Description: The Baseline Hb was defined as the average of the last 2 central laboratory Hb values taken on or prior to the first dose date. The average for the PEP was calculated as the average of all Hb measurements from the central laboratory within the three visit windows during Weeks 20 through 26, regardless of intercurrent events. Analysis was conducted using an analysis of covariance (ANCOVA) model with multiple imputation for missing data with randomization stratification factors and Baseline Hb as covariates. Change from Baseline was calculated as PEP value minus the Baseline value.
Time Frame: Baseline; Weeks 20 to 26
Population: Randomized Population
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Vadadustat QD | Vadadustat TIW | Darbepoetin Alfa
Number analyzed (Participants) | 105 | 106 | 108
Grams per deciliter (g/dL) | 0.07 (0.12) | -0.19 (0.12) | 0.34 (0.12)

2. Secondary Outcome: Change From Baseline in Hb to the Average Over the Secondary Evaluation Period (SEP) (Weeks 46 to 52)
Description: The Baseline Hb was defined as the average of the last 2 central laboratory Hb values taken on or prior to the first dose date. The average for the SEP was calculated as the average of all Hb measurements from the central laboratory within the three visit windows during Weeks 46 through 52, regardless of intercurrent events. Analysis was conducted using an ANCOVA model with multiple imputation for missing data with randomization stratification factors and Baseline Hb as covariates. Change from Baseline was calculated as SEP value minus the Baseline value.
Time Frame: Baseline; Weeks 46 to 52
Population: Randomized Population
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Vadadustat QD | Vadadustat TIW | Darbepoetin Alfa
Number analyzed (Participants) | 105 | 106 | 108
g/dL | 0.04 (0.15) | 0.03 (0.15) | 0.44 (0.15)

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to Week 56 (from first dose of study drug to last dose + 4 weeks of follow-up)
Description: All serious and non-serious adverse events were collected in the Safety Population which consisted of all participants in the randomized population who received at least 1 dose of study drug. Participants received treatment per dosing schedule and the data was not collected for each dose level separately.
Arm/Group | Vadadustat QD | Vadadustat TIW | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 12/105 | 9/104 | 7/108
Serious Adverse Events (participants affected / at risk) | 47/105 | 47/104 | 47/108
Other Adverse Events (participants affected / at risk) | 46/105 | 49/104 | 46/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat QD (N=105) | Vadadustat TIW (N=104) | Darbepoetin Alfa (N=108)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 5
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 6 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 3 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0
Parathyroid hyperplasia (Endocrine disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 2
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 2 | 4
COVID-19 pneumonia (Infections and infestations) | 7 | 8 | 4
Candida pneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 2
Cryptococcal fungaemia (Infections and infestations) | 1 | 0 | 0
Device related bacteraemia (Infections and infestations) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 2
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 1 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 1 | 2
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 2
Muscle abscess (Infections and infestations) | 0 | 1 | 0
Necrotising soft tissue infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1 | 2
Otitis media staphylococcal (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 0
SARS-CoV-2 sepsis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 3
Septic shock (Infections and infestations) | 1 | 1 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vascular graft infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 2 | 3
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 4 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 2 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0
Steal syndrome (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat QD (N=105) | Vadadustat TIW (N=104) | Darbepoetin Alfa (N=108)
Anaemia (Blood and lymphatic system disorders) | 5 | 7 | 7
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 14 | 15 | 6
Nausea (Gastrointestinal disorders) | 12 | 6 | 6
Vomiting (Gastrointestinal disorders) | 10 | 4 | 6
Oedema peripheral (General disorders) | 6 | 0 | 3
COVID-19 (Infections and infestations) | 12 | 11 | 10
Fall (Injury, poisoning and procedural complications) | 10 | 6 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 5 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2
Hypertension (Vascular disorders) | 6 | 11 | 10

LIMITATIONS AND CAVEATS:
Per the protocol, data was collected by the arm to which participants were randomized and not by dose received in vadadustat QD or vadadustat TIW arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT04313153/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04313153/SAP_001.pdf